CLINICAL TRIAL: NCT05937919
Title: CLDN18.2 Targeted 68Ga-PMD22 PET Imaging in Patients With Gastrointestinal Tumours
Brief Title: 68Ga-PMD22 PET/CT Examination Targeting CLDN18.2
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-PMD22
Record Dates: First submitted 2023-06-19; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Gastrointestinal Cancer
Keywords: CLDN18.2; Gastric Cancer; Colorectal Cancer; Positron emission tomography
MeSH Terms: conditions — Gastrointestinal Neoplasms; Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-PMD22 PET/CT dynamic scan (Experimental): 68Ga-PMD22 PET/CT scan Dosimetry study about 6 patients were injected with 2-4 (MBq) per kilogram body weight of 68Ga-PMD22 PET/CT in one dose intravenously and underwent wholebody scan at 5min#15min#30min#60min#90min#120min#180min, then analysis of dosimetric distribution of radiopharmaceuticals in human body by HERMES software.
  Interventions: Drug: Intravenous injection of 68Ga-PMD22
- 68Ga-PMD22 PET/CT scan at one time (Experimental): After the dynamic scan completed, choose an optimal imaging examination time for PET examination of other patients.
  Interventions: Drug: Intravenous injection of 68Ga-PMD22

INTERVENTIONS:
Drug: Intravenous injection of 68Ga-PMD22 — 68Ga-PMD22 were intravenous injected into the patients before PET/CT scans
  Other Names: 68Ga-PMD22

SUMMARY:
To investigate the ability of the CLDN18.2-targeted 68Ga-PMD22 tracer to detect CLDN18.2 expression in patients with gastric and colorectal cancer and other gastrointestinal tumours.

DETAILED DESCRIPTION:
The 2016 FAST study brought a "new star" target for gastric cancer - CLDN18.2 (claudin 18 splice variant 2,CLDN18.2), which belongs to the CLDN family of tight junction proteins and is involved in the formation of paracellular tight junctions and maintenance of cell polarity. CLDN18.2 is mainly found in the normal gastric mucosa (normal gastric glands, principal cells, mural cells, endocrine cells) where the differentiation cycle is short and renewal is rapid, and in the duodenal panniculocytes, but not in the gastric stem cell region. It is now generally accepted that CLDN18.2 is expressed in normal gastric tissue confined to the tight junctions at the outer base of the gastric mucosal cells, whereas tumours undergo a change in cell polarity during malignant transformation, resulting in widespread exposure of CLDN18.2 to the cell membrane surface. The CLDN18.2 gene is also aberrantly activated and highly specific and stably expressed in specific tumour tissues, participating in the proliferation, differentiation and migration of tumour cells, making it a potentially effective target for anti-tumour drugs.

In this study, a molecular probe PMD22 targeting CLDN18.2 was synthesised in a previous study and a 68Ga-PMD22 injection was developed for clinical trials. The preliminary study showed that the tracer has good safety and good imaging effect. It is proposed to further conduct exploratory PET/CT imaging studies on patients with gastric cancer, colorectal cancer and other gastrointestinal tumours, to provide a new technique for in vivo, non-invasive and visual detection of CLDN18.2 expression level and spatial distribution for patients with gastric cancer, colorectal cancer and other gastrointestinal tumours, and to validate its clinical application value for the diagnosis of gastric cancer, colorectal cancer and other gastrointestinal tumours.

ELIGIBILITY:
Inclusion Criteria:

* In the near future (within 2 months), patients who plan to undergo puncture biopsy or undergo tumor surgical treatment or are clinically highly suspected of cancer (including primary and tumor recurrence and metastasis)
* Able to understand and voluntarily sign informed consent forms, with good compliance

Exclusion Criteria:

* Severe abnormalities in liver and kidney function
* Suffering from claustrophobia or other mental illnesses
* Pregnant and lactating women

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-28 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Dosimetric distribution of radiopharmaceuticals | 2 months
  Input the 68Ga-PMD22 PET data of 5-6 patients into HERMES software, and analyze the dose distribution of radioactive drugs in human body through HERMES software
Standardized uptake value | 2 months
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in breast tumor will be measured. SUV were obtained by a self-made software and referring to phantom study.If the SUV value cannot be obtained, the COUNTS of target organ/background ratio between the lesion and surrounding tissues shall be used for calculation.

SECONDARY OUTCOMES:
Number of participants with drug-related adverse events | 1 month
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed by phone call and assessed the safety of 68Ga-PMD22, including blood pressure, blood function, liver and kidney function data, gastrointestinal reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, China

REFERENCES:
- [Derived] Wang R, Bai Z, Zhong W, Li C, Wang J, Xiang J, Du J, Jia B, Zhu Z. Synthesis, preclinical evaluation and pilot clinical translation of [68Ga]Ga-PMD22, a novel nanobody PET probe targeting CLDN18.2 of gastrointestinal cancer. Eur J Nucl Med Mol Imaging. 2024 Oct;51(12):3731-3743. doi: 10.1007/s00259-024-06808-5. Epub 2024 Jun 27. PMID 38926162